CLINICAL TRIAL: NCT02035150
Title: The Effect of Ingesting Breakfasts Varying in Fiber on Appetite and Weight Change in Overweight Subjects
Brief Title: Effect of Different Fiber Breakfasts on Appetite and Weight Change in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Obesity and Nutrition Research Center (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Principal Investigator, Dr. Allan Geliebter, Research Scientist, New York Obesity and Nutrition Research Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 98-022
Record Dates: First submitted 2014-01-08; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: breakfast; oatmeal; appetite; cholesterol
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oatmeal Breakfast (Experimental): Participants will consume oatmeal breakfast daily for 4 weeks
  Interventions: Dietary Supplement: Oatmeal
- Frosted Flakes (Experimental): Participants will consume a frosted flakes breakfast daily for 4-weeks
  Interventions: Dietary Supplement: Frosted Flakes
- No Breakfast (Placebo Comparator): Participants will consume no breakfast for a 4-week period
  Interventions: Dietary Supplement: No Breakfast

INTERVENTIONS:
Dietary Supplement: Oatmeal — A breakfast consisting of oatmeal
  Other Names: Quaker Quick Oats
  Arms: Oatmeal Breakfast
Dietary Supplement: Frosted Flakes — A breakfast consisting of Frosted Flakes and milk
  Other Names: Kelloggs Frosted Flakes
  Arms: Frosted Flakes
Dietary Supplement: No Breakfast — A breakfast consisting of plain water
  Arms: No Breakfast

SUMMARY:
Regular breakfast consumption may help lower body weight reduce body fatness and improve cardiovascular disease risk factors. However, the best kind of breakfast to consume to achieve these effects is unclear. We hypothesized that a high fiber breakfast would suppress appetite, lower body weight and improve cardiovascular disease risk factors compared with a no-fiber breakfast.

DETAILED DESCRIPTION:
Participants will report to the hospital cafeteria between 0800 and 0900h following an overnight fast every weekday for 4 consecutive weeks. On arrival, participants will be provided will the allocated breakfast and will be given 15 min to consume all the foods provided. The oatmeal breakfast will consist of 80g dry oatmeal (Quaker Quick Oats) prepared with 120mL fat-free milk and 230mL water. The frosted flakes breakfast will consist of 62g frosted flakes and 160mL whole milk and 190mL water served on the side. The No-breakfast (control) will consist of only 350mL plain water. All participants will also receive 200mL decaffeinated coffee with 12mL non-dairy creamer and 1g packet of non-caloric sweetener. On Friday of each week participants will be provided with two portions of the breakfasts to take home at consume on the weekend days. On the first day of the intervention and weekly thereafter participants will complete 3hr subjective appetite ratings responses to the breakfast. Laboratory assessments including body weight, composition, blood pressure and a fasting blood sample will be collected before the start of the intervention and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI >27kg/m2
* Weight stable (<5% weight change in past 3 months)

Exclusion Criteria:

* Smokers
* Regular use of medications
* Currently undertaking a weight-loss or exercise program
* Females who are pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1998-03; Primary Completion 2000-02 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Change in body weight over 4 week intervention
  Body weight will be measured at baseline and following 4-week breakfast intervention

SECONDARY OUTCOMES:
Subjective appetite | Appetite ratings in response to breakfast will be collected for 3hs on the first day of the study and after 1, 2, 3 and 4 weeks of the intervention
  Ratings of hunger and Fullness will be collected on a 6 point rating scale with 0 labelled not at all, 40 moderately, 60 quite, 80 very and 100 extremely.
Change in plasma metabolic risk factors | At baseline and following 4-week intervention
  A fasting blood sample will be collected and analyzed for glucose, insulin, triacylglycerol, leptin and cholesterol
Resting Energy Expenditure | Resting energy expenditure will be measured at baseline and following the 4 week intervention
  Resting energy expenditure measurements will be collected whilst subjects are fasting, resting in a semi-supine position under thermoneutral conditions with a ventilated hood and metabolic cart.

OTHER OUTCOMES:
Blood pressure | At baseline and following 4-week intervention
  Systolic and diastolic blood pressure will be measured at baseline and following 4-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — New York Obesity Nutrition Research Center